CLINICAL TRIAL: NCT03949725
Title: Evaluating the Hans Kai Program for Canadian Adults Via an 18-month Mixed Methods Randomized Controlled Trial
Brief Title: A Mixed Methods Randomized Controlled Trial Evaluating the Hans Kai Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: NorWest Co-op Community Health (Other)
Responsible Party: Principal Investigator, Dylan MacKay, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS21887 (H2018:241)
Record Dates: First submitted 2019-05-08; First posted 2019-05-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Mental Health; Social Isolation; Loneliness; Health-Related Behavior
Keywords: Health Promotion; Peer-led; Mixed Methods RCT
MeSH Terms: conditions — Psychological Well-Being; Social Isolation; Health Behavior

STUDY DESIGN:
Intervention Model Description: The intervention study model is a 2-arm randomized control trial with a 2:1 allocation of participants to the treatment condition (i.e., the Hans Kai program) or the control condition (i.e., usual care without the Hans Kai program). After 6 months in the control condition, participants in the control group will join the Hans Kai program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hans Kai program (Experimental): The Hans Kai program is a peer-led, preventative, self-sustaining, community-based health promotion program for adults of all ages, genders, and socioeconomic circumstances who wish to maintain or improve their health. Hans Kai empowers individuals to take control of their own health and provides a unique opportunity for participants to have an active role in improving or maintaining their health and wellbeing.
  Interventions: Behavioral: Hans Kai Program
- Wait list control (No Intervention): Participants in the waitlist control group will remain as close to a 'typical' community member as possible as they will be able to receive any health programming normally available to them in Winnipeg, except the Hans Kai program. Standard of care is made available to all members of the control group as related to the healthcare rights of Canadians and Manitobans holding a Manitoba health card. NorWest staff will provide support to the community members without a Manitoba health card in obtaining one. The only deviation from standard care in the waitlist control group will be the pre- and post-intervention visits during which the control participants will fill out self-report questionnaires and undergo physical assessments.

INTERVENTIONS:
Behavioral: Hans Kai Program — In Hans Kai, first, participants attend a 2-month Health School to develop the skills necessary to improve their health and wellbeing. The Health School includes sessions on health indicators; nutrition, grocery shopping and meal planning; physical activity; stress, coping, and health (sleep); and primary care through the years. After participants complete the Health School, they form Hans Kai groups (of 3 or more adults) and begin to meet regularly (at least once a month) independently of facilitators, in a self-sustaining model.
  Arms: Hans Kai program

SUMMARY:
The Hans Kai trial is a mixed methods randomized controlled trial evaluating the effectiveness of the peer-led health promotion Hans Kai program for Canadian adults with or without chronic health conditions. The Hans Kai trial also aims to identify the strengths and weaknesses of the Hans Kai program as well as the facilitators and barriers to its implementation from the perspectives of the program participants and facilitators. The intervention (Hans Kai program) consists of an 8-week health school that program participants attend to develop health knowledge and skills. Next, program participants form Hans Kai groups of 3 or more people, who meet on a monthly basis independently in a peer-led self-sustaining model. The trial will measure the impact of Hans Kai, compared to waitlist control, on program participants' mental health; social connections; health-related knowledge and empowerment (i.e., self-efficacy and self-determination); health-promoting behaviors (i.e., diet, alcohol consumption, tobacco use, physical activity, and sleep); and clinical measures of cardio-metabolic health.

DETAILED DESCRIPTION:
The Hans Kai trial will follow a prospective mixed methods intervention design involving an RCT and an interpretative descriptive qualitative study. The mixed methods intervention design is a mixed methods approach to research in which the collection, analysis, and integration of both quantitative and qualitative data are embedded within an experimental quantitative research design. The objective of gathering qualitative data within an experiment, along with the quantitative data on the outcome measures, is to gain an understanding of the personal, contextual experiences of the study participants.

In this mixed methods intervention study design, quantitative data on the outcomes of interest will be collected along with qualitative data on the experiences of program participants and facilitators, and integrated within an intervention trial (i.e., RCT) to address the research objectives (see next section for details). The primary research design in this study will be a quantitative intervention trial or RCT that will follow a pragmatic randomized wait-list-control design with an 18-month follow-up. The RCT will involve the collection, analysis, and interpretation of quantitative data (self-reports and objective indicators) on primary, secondary, and tertiary outcomes that will be gathered to evaluate the effectiveness of the Hans Kai program in promoting the health and wellbeing of Canadian adults. To enrich the RCT results, the secondary qualitative strand of the study will be added during and after the intervention by embedding a combination of convergent and explanatory sequential designs into the RCT.

ELIGIBILITY:
Inclusion Criteria. Participants may enter the trial if all the following apply.

* Age 18 years or above.
* Any gender.
* Willingness and ability to give informed consent for participation in the trial.
* Ability to speak and read English at a grade 6 level.
* Motivation to make a lifestyle change as indicated on the research study consent form.
* Stable health status that allows participation in the group context, including performing light exercise, to be determined by the participant and study Hans Kai staff.
* Ability and willingness to comply with all trial requirements, to be determined by the research team.

Exclusion Criteria. Participants may not enter the trial if any of the following apply.

* Age under 18 years.
* Cognitive impairment that prevents the person from providing informed consent or participating in the program.
* Existing relationship with the research team, such as supervisory relationship (e.g., student or employee) or familial relationship (e.g., child or spouse).
* Frailty that prevents the person from participating in group activities or exercise.
* Participation in another research trial in the past 12 weeks.
* Unstable health or serious illness, for example, dementia, terminal illness, or recent significant medical diagnosis.
* Inability to attend the scheduled Hans Kai Health School and assessment sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Mental Health | 6 months
  Mental health will be measured using the Mental Health Continuum Short Form (MHC-SF). The MHC-SF is a standardized self-report questionnaire that measures emotional, social, and psychological well-being by assessing the regularity with which respondents experience symptoms of positive mental health. The questionnaire includes 14 items asking respondents to indicate on a 6-point Likert scale (ranging from 0 = never to 5 = everyday) how often in the previous month they experienced symptoms of emotional, social, and psychological wellbeing. Item responses are summed, yielding a total score ranging from 0 to 70, with higher scores indicating more positive wellbeing.

SECONDARY OUTCOMES:
Social Connectivity | 6 months
  Feelings of loneliness and social isolation will be measured using the revised UCLA Loneliness Scale. This is a standardized 20-item scale designed to measure one's subjective feelings of loneliness and social isolation by asking respondents to rate each item on a scale from 1 (Never) to 4 (Often). Single-item scores are summed to obtain a total score ranging from 20 to 80, with lower scores indicating greater loneliness and/or social isolation.
Health-related Knowledge and Empowerment | 6 months
  Health-related knowledge and empowerment in the form of self-efficacy and self-determination will be measured using the Perceived Health Competence Scale (PHCS). This is a standardized measure of general health management self-efficacy beliefs designed to assess respondents' self-perceived ability to accomplish health-related goals and manage their health positively. The 8 items ask respondents to rate on a 5-point Likert scale ranging from 1 = strongly disagree to 5 = strongly agree the degree to which they feel capable of effectively managing their health outcomes. Single item scores are summed to create an overall score ranging from 8 to 40, with higher scores indicating a higher self-perceived health competence.
Diet, Alcohol Consumption, & Tobacco Use | 6 months
  Changes in nutritional behavior (diet), alcohol consumption, and tobacco use will be measured using a modified version of the Healthy Eating Assessment. The adapted self-report scale includes a total of 22 items divided into two main sections: (1) a first section that includes 18 items evaluating respondents' eating habits, and (2) a second section including four items that assess respondents' alcohol consumption and tobacco use.
Sleep Quality, Habits, and Patterns | 6 months
  The standardized self-report questionnaire Pittsburgh Sleep Quality Index (PSQI) will be used to subjectively measure sleep quality, habits, and patterns. This scale includes nine items that assess seven aspects of sleep: (1) subjective sleep quality; (2) sleep latency; (3) sleep duration; (4) habitual sleep efficiency; (5) sleep disturbances; (6) use of sleeping medications; and (7) daytime dysfunction over the last month. Scoring varies across items; however, an overall score can be calculated by summing the seven component scores, yielding a Global PSQI score ranging from 0 to 45, with higher scores indicating poorer sleep quality. Sleep quality and patterns will also be measured objectively using data provided by the Fitbits that participants will wear for a week at each assessment point. The average of these seven measurements will be used as an indicator of sleep patterns and quality
Physical Activity: Moderate-to-Vigorous Physical Activity (MVPA) | 6 months
  Physical activity levels will be measured by recording the minutes of moderate-to-vigorous physical activity (MVPA) study participants engage in each day over a 7-day period using a Fitbit that study participants will wear for 1 week. The average of these seven measurements will be used as an indicator of participants' level of physical activity.
Physical Activity: Step Count | 6 months
  At each assessment point, a daily step count will be recorded over a 7-day period. The average of these seven measurements will be used as an indicator of participants' level of physical activity at that timepoint of data collection.

OTHER OUTCOMES:
Waist Circumference | 6 months
  Waist circumference in cm will be measured in triplicate, to the nearest 0.1 cm at the umbilicus, between the last rib and the iliac crest using a fibreglass tape measure by a registered nurse.
Systolic Blood Pressure | 6 months
  Systolic blood pressure in mmHg will be measured in triplicate, on the non-dominant arm in a sitting position by a registered nurse using a validated oscillometric blood pressure monitor.
Diastolic Blood Pressure | 6 months
  Diastolic blood pressure in mmHg will be measured in triplicate, on the non-dominant arm in a sitting position by a registered nurse using a validated oscillometric blood pressure monitor.
Fasting Blood Sugar | 6 months
  Blood glucose will be measured in mmol/L by finger stick capillary blood sampling using a calibrated glucometer.
Heart Rate | 6 months
  Heart Rate in beats per minute will be measured in triplicate, on the non-dominant arm in a sitting position by a registered nurse using a validated oscillometric blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Mackay, Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- NorWest Co-op Community Health, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
Following deidentification, all of the individual participant data (IPD) collected during the trial will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will be available beginning immediately following publication and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal and whose proposed use of the data has been approved by the trial PI.

REFERENCES:
- [Derived] Cameranesi M, Mollard R, Balshaw R, MacKay D. The Hans Kai trial: study protocol of a mixed methods randomized controlled trial evaluating a peer-led health promotion program for adults with or without noncommunicable diseases. Trials. 2023 Oct 24;24(1):689. doi: 10.1186/s13063-023-07708-z. PMID 37875962